CLINICAL TRIAL: NCT03667846
Title: Leveraging Biomarkers for Personalized Treatment of Alcohol Use Disorder Comorbid With Post Traumatic Stress Disorder
Brief Title: Leveraging Biomarkers for Personalized Treatment of Alcohol Use Disorder Comorbid With PTSD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-01405; P01AA027057 (NIH)
Record Dates: First submitted 2018-08-22; First posted 2018-09-12 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Post Traumatic Stress Disorder; Alcohol Use Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcoholism | interventions — Topiramate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo
- Topiramate (Experimental): Week 0-1: 25 mg qhs Week 1-2: 25 mg qAM, 25 mg qhs Week 2-3: 25 mg qAM, 50 mg qhs Week 3-4: 50 mg qAM, 50 mg qhs Week 4-5: 50 mg qAM, 75 mg qhs Week 5-6: 75 mg qAM, 75 mg qhs Week 6-7: 75 mg qAM, 100 mg qhs Week 7-8: 100 mg qAM, 100 mg qhs Week 8-10: 100 mg qAM, 100 mg qhs Week 10-12: 100 mg qAM, 100 mg qhs Week 12-14: 2-week taper
  Interventions: Drug: Topiramate

INTERVENTIONS:
Drug: Topiramate — Generic topiramate, FDA-approve for clinical use, will be purchased in 25mg, 50mg, and 100mg strengths, and encapsulated.
  Other Names: Topamax
  Arms: Topiramate
Other: Placebo — Placebo tablets will be encapsulated in identical capsules.
  Arms: Placebo

SUMMARY:
This is a double-blind, 2-group randomized controlled trial evaluating the effects of topiramate versus placebo in patients with comorbid PTSD and moderate-to-severe AUD. This trial will provide one of the first rigorous tests of whether the effects of topiramate in AUD generalize to patients with co-occurring PTSD, and one of the first rigorous tests of whether topiramate has beneficial effects on PTSD symptoms in this population. It will be the first study to test whether the rs2832407 genotype predicts clinical response to topiramate for AUD and PTSD in patients with both disorders. Further, it will contribute to the understanding of topiramate's mechanisms of action in the co-morbid AUD/PTSD population, and to the discovery of predictors of treatment response.

DETAILED DESCRIPTION:
Alcohol use disorder (AUD) and post-traumatic stress disorder (PTSD) are highly comorbid, and present a clinical challenge for which existing treatments have limited efficacy. Existing clinical evidence suggests treatments that simultaneously address symptoms of both PTSD and AUD should be more efficacious than treating either disorder in isolation. The overlap in the neurobiological basis of PTSD and AUD (involving alterations in incentive salience, stress/negative affect, and executive control network functioning) suggests that there could be treatments that would effectively treat both disorders. However, there is no pharmacotherapy or psychotherapy treatment that is clearly effective for both disorders.

Topiramate, an FDA-approved anticonvulsant with effects on GABAergic and glutamatergic signaling, has demonstrated efficacy in the treatment of AUD in several randomized clinical trials (RCTs), and has also been tested in several open-label and small RCTs for treatment of PTSD with some evidence of effectiveness. Positive results in one open-label trial and one small RCT in patients with co-occurring PTSD and AUD suggest that topiramate may have beneficial effects on symptoms of both PTSD and AUD in this population. Preclinical work also supports the efficacy of topiramate in ameliorating anxiety-like behavior and altered stress response in animal models of stress and chronic alcohol exposure. A recent clinical study demonstrated that the effects of topiramate on alcohol use were moderated by a polymorphism of the GRIK1 gene (coding for the kainate receptor GluK1 subunit), such that significant benefit was found only among rs2832407 C-allele homozygotes.

This trial is designed to contrast acute and persisting effects of topiramate to those of placebo treatment in a sample of 150 participants with comorbid PTSD and moderate to severe AUD, and to evaluate the moderating effect of rs2832407 genotype on medication effects. Drug will be titrated over 8 weeks to a maximum dose of 200 mg and continued for 4 more weeks for a total of 12 weeks of treatment, followed by a 2-week taper. Alcohol and PTSD-related outcomes will be assessed at multiple time points throughout the study. Plasma biomarkers and neuropsychological assessments will be obtained at baseline and at week 12. In support of the overall aims of the center focusing on personalized medicine, the trial will serve as a platform for studies of topiramate's effects on brain chemistry and function as measured by fMRI, and EEG . Data from this clinical trial will also contribute to Overall Center Aims investigating the relationship of plasma biomarkers to neuroimaging markers.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 18-70 years old
2. DSM-5 diagnosis of moderate or severe AUD (using SCID5)
3. Endorse a desire to cut down or stop drinking
4. At least 4 heavy drinking days (4 or more drinks per day for a woman, 5 or more drinks per day for a man) in the 30 days prior to screen
5. DSM-5 current diagnosis of PTSD with the Clinician Administered PTSD Scale OR subPTSD diagnosis (meeting criterion A, F, G, H and at least 6 symptoms across any criteria B-E) with Clinician Administered PTSD Scale (CAPS-5)
6. If of childbearing potential (male or female), are willing to use contraception for duration of the trial
7. Able to provide at least 2 locators
8. Able to provide voluntary informed consent
9. Confirms they are reliably domiciled

Exclusion Criteria:

1. Current alcohol withdrawal (CIWA-Ar score >7)
2. DSM-5 diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder I, current significant suicidality (assessed using the C-SSRS), any significant suicidal behavior in the past 12 months, or any history of serious suicide attempts requiring hospitalization, or active homicidality
3. DSM-5 diagnosis of current severe substance use disorder for a substance other than alcohol or nicotine
4. Any history of severe traumatic brain injury (assessed using the OSU TBI-ID modified). If current (past 12 months) mild/moderate TBI and CSI score ≥12 (for either lifetime month or current month), the PI will determine eligibility.
5. Exposure to trauma in the last 30 days, including police duty or military service
6. Significantly impaired liver function defined as a) alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 5 x upper limit of normal (ULN); b) ALT or AST > 3 x ULN with concomitant total bilirubin > 2.0 x ULN; or c) ALT or AST ≥ 3 x ULN with the appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia
7. Other medical conditions which would preclude safe participation in the study
8. Significant laboratory abnormalities, including significantly impaired hepatic function, abnormalities in complete blood count or metabolic panel
9. Current use of medications with the potential for adverse drug-drug interactions including but not limited to CNS depressants specified anticonvulsants (such as: Phenytoin, Carbamazepine and Depakote), metformin, and pharmacologic treatments for addictions including alcohol use disorder ,and other Carbonic Anhydrase inhibitors (i.e. zonisamide, acetazolamide, dichlorphenamide). Oral contraceptives are permitted as long as participants who are on an estrogen and/or estrogen-progesterone form use a double barrier contraceptive. Antidepressant medications are permitted if participants have been on a stable dose for at least 4 weeks prior to screening and the dose may not be changed during treatment phase (weeks 0-14) of the study.
10. Pregnancy or lactation
11. Current treatment for AUD (with the exception of AA/12-step treatment and/or psychosocial treatment initiated more than 2 months prior to the screening visit)
12. Current treatment for methadone or opioid abuse
13. Psychotherapy for PTSD or other psychiatric condition, if initiated within 3 months of screening
14. Allergy or hypersensitivity to topiramate
15. Active legal problems likely to result in incarceration within 12 weeks of treatment initiation
16. Significantly impaired renal function defined as) creatinine clearance rate <70 mL/min/1.73 m2.
17. High risk of adverse emotional or behavioral reaction, and/or an inability to understand study procedures or the informed consent process, based on investigator's clinical evaluation (e.g., evidence of serious personality disorder, antisocial behavior, serious current stressors, lack of meaningful social support)
18. Inpatient psychiatric treatment in the last 12 months, with the exception of detox and extended Emergency Department stays

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-10-10 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Measure of Time-line Follow-back (TLFB) | Day 1
  Retrospective estimate of daily alcohol consumption over a time period ranging from 7 days to 24 months prior to initial interview
Percent Day Abstinent from Alcohol | Week 9 to Week 12
  Percentage of day abstinent from alcohol between week 9 and week 12
PCL-5 score | Week 9 to Week 12
  20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. The symptom severity score (range - 0-80) can be obtained by summing the scores for each of the 20 items. Each question is measured on a 5-point Likert (0 = "Not at all" to 4 = "Extremely"). A total symptom severity score (range - 0-80; 80 being more severe) can be obtained by summing the scores for each of the 20 items.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Marmar, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be made available within twelve months of database lock or following publication of primary manuscript, whichever occurs first. Data will be available indefinitely.
Access Criteria: Anyone who wishes to access the data.